CLINICAL TRIAL: NCT06460077
Title: Exploring Pathology Related to Slowly Expanding Lesions Using Advanced Imaging
Acronym: SELPET
Status: Enrolling by invitation | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SELPET
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Multiple Sclerosis: Patients who have previously participated in PET-imaging studies and from whom slowly expanding lesions as well as TSPO-rim-positive lesions and iron rims at the edge of lesions are found

SUMMARY:
This is an open, follow-up study to compare the performance of three critical imaging methods to detect chronic active lesions in Multiple Sclerosis (MS) in vivo.

DETAILED DESCRIPTION:
Smoldering inflammation is recognized as a critical contributor to MS progression-related central nervous system (CNS) damage. Activated microglia and macrophages particularly at chronic lesion edge are believed to promote lesion growth. Reversing their harmful activity may prove to be an efficient way to halt progression independent of relapses in MS.

These smoldering, or chronic active lesions can be detected in vivo using advanced imaging techniques. 1) Specific algorithms can be used to identify lesion growth, with a hypothesis that the slowly evolving lesions (SEL) are the ones harboring a rim of activated microglial cells, which contribute to damage in the surrounding tissue, and lesion growth. 2) Lesions partially or entirely surrounded by rims of increased tissue intensity on QSM-MRI (quantitative susceptibility mapping) sequences are considered as iron rim lesions, with iron-containing proinflammatory microglia/macrophages at the lesion edge. 3) In addition, 18 kDa translocator protein-positron emission tomography (TSPO-PET) imaging can be used to identify chronic active lesions based on TSPO-expression by activated innate immune cells, and their gathering at the edges of chronic active lesions. The TSPO-PET analysis of chronic active lesions can be semi-automated, and the specific radioligand binding at the chronic active lesion edge can be quantitated, which enhances the sensitivity of this method.

Despite existing preliminary data demonstrating increased QSM signal TSPO-positive lesions, it is yet to be demonstrated how these three imaging methods perform in identifying chronic active lesions when compared to each other at larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent form
* MS diagnosis in accordance with McDonald 2017 criteria
* Available longitudinal brain MR images (minimum 1 year)
* Simultaneous QSM MRI sequence and TSPO-PET
* Lesions with iron rim/s

Exclusion Criteria:

* Patients with other neurodegenerative disease than MS
* Patients with other autoimmune disease than MS
* Patients with other significant or malignant underlying disease of any other organ system
* Patients that are pregnant or breast-feeding
* Corticosteroid treatment within 4 weeks of imaging
* Patients with significant abnormal findings other than MS in the screening MRI
* Patients with claustrophobia, or a history of moderate to severe anxiety disorder or panic attacks (which could potentially lead to preterm termination of the imaging)
* Contraindication to PET scan investigations
* Exposure to experimental radiation in the past 12 months such that radiodosimetry limits would be exceeded by participating in this study
* Intolerance to previous PET scans; i.e. previous hypersensitivity reactions to any PET ligand or imaging agent or failure to participate in and comply with previous PET scans

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 52 MS patients with simultaneous QSM-MRI and TSPO-PET and with available longitudinal brain MRI images (minimum 1 year) have been identified. With an average detection frequency of >= 1 SEL in 70% of MS patients, there will be sufficient imaging material for successful conduct of the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of lesions | 18 months, 36 months
  The number of lesions identified using each respective method
Co-localization of lesions | 18 months, 36 months
  Potential co-localization of the RIM+ lesions identified using the various methods.

SECONDARY OUTCOMES:
Correlation of PET imaging and clinical variables | 18 months, 36 months
  Imaging variables from PET imaging correlated with clinical status of the patient evaluated with Expanded Disability Status scale (EDSS). EDSS describes the disability level and ranges from 0 to 10, where 0 means no disability due to MS and 10 means death due MS.
Correlation of magnetic resonance imaging and clinical variables | 18 months, 36 months
  Imaging variables from MR imaging correlated with clinical status of the patient evaluated with Expanded Disability Status scale (EDSS). EDSS describes the disability level and ranges from 0 to 10, where 0 means no disability due to MS and 10 means death due MS.
Correlation of quality of life questionnaires and clinical variables | 18 months, 36 months
  Correlation of quality of life questionnaires and clinical status of the patient evaluated with Expanded Disability Status scale (EDSS). EDSS describes the disability level and ranges from 0 to 10, where 0 means no disability due to MS and 10 means death due MS.
Correlation of neuropsychological evaluation and clinical variables | 18 months, 36 months
  Correlation of neuropsychological evaluation and clinical status of the patient evaluated with Expanded Disability Status scale (EDSS). EDSS describes the disability level and ranges from 0 to 10, where 0 means no disability due to MS and 10 means death due MS.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, MD,Professor, Principal Investigator — Turku University Hospital, division of clinical neurosciences
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland